CLINICAL TRIAL: NCT06104306
Title: A Phase 4 Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Oral B/F/TAF After Discontinuing Injectable CAB + RPV
Brief Title: Study of B/F/TAF in Participants Switching From CAB + RPV to B/F/TAF for HIV-1 Infection (EMPOWER)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-380-6738; 2023-506660-13 (Other: European Medicines Agency)
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- B/F/TAF (Experimental): Participants will receive a fixed dose combination of B/F/TAF 50/200/25 mg once daily for 24 weeks.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — Tablets administered orally without regard to food
  Other Names: Biktarvy ®

SUMMARY:
The goal of this clinical study is to learn how safe it is to switch to an oral therapy of Bictegravir/Emtricitabine/Tenofovir (B/F/TAF) from Cabotegravir + Rilpivirine (CAB+RPV) in participants living with virologically suppressed human immunodeficiency virus type 1 (HIV-1), meaning participants with HIV RNA levels below detectable levels.

The primary objective of this study is to assess the safety of switching to B/F/TAF in virologically suppressed participants unable/unwilling to continue on CAB+RPV intramuscular (IM) injections or wishing to switch to oral therapy through Week 12.

ELIGIBILITY:
Key Inclusion Criteria:

* People with human immunodeficiency virus type 1 (HIV-1) (PWH) or provider decision to switch off cabotegravir + rilpivirine (CAB+RPV) intramuscular (IM) injections due to intolerance, inconvenience, adverse events (AEs), or willing to switch to (and intention to remain on) daily bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF).
* Currently virologically suppressed (HIV-1 ribonucleic acid (RNA) < 50 copies/mL) on CAB+RPV IM injections every 2 months.
* Currently on CAB+RPV IM injections every 2 months and received at least one dose of CAB+RPV IM injection; no missed CAB+RPV injections.
* Ability to receive B/F/TAF up to 7 days prior to the next scheduled dose of CAB+RPV.
* Documented plasma HIV-1 RNA < 50 copies/mL during treatment for ≥ 6 months preceding the screening visit.
* No documented or suspected resistance to bictegravir, emtricitabine, or tenofovir.

Key Exclusion Criteria:

* History of B/F/TAF intolerance.
* History of previous integrase strand-transfer inhibitor (INSTI) virologic failure including CAB+RPV.
* Requirement for ongoing therapy with any prohibited medications listed in local prescribing information for B/F/TAF starting within 30 days prior to screening until 30 days following the last dose of study drug.
* Have been treated within 3 months of study screening or expected to receive during the study immunosuppressant therapies or chemotherapeutic agents (eg, chronic (at least 4 weeks) systemic steroids, immunoglobulins, and other immune- or cytokine-based therapies)
* Need for oral antiretroviral therapy (ART) bridge or use of other antiretroviral (ARV) agents prior to starting B/F/TAF on Day 1

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- United States (10):
  - Franco Felizarta, MD, Bakersfield, California
  - BIOS Clinical Research, Palm Springs, California
  - UC San Diego AntiViral Research Center (AVRC), San Diego, California
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Bliss Health, Orlando, Florida
  - Indiana University Infectious Diseases Research, Indianapolis, Indiana
  - Boston Medical Center, Boston, Massachusetts
  - Las Vegas Research Center, Las Vegas, Nevada
  - Saint Michael's Medical Center, Newark, New Jersey
  - MultiCare Rockwood Main Clinic, Spokane, Washington
- Canada (3):
  - Hamilton Health Sciences-SIS Clinic, Hamilton
  - St. Michael's Hospital, Toronto
  - University Health Network - Toronto General Hospital, Toronto
- France (5):
  - CHU Bordeaux - Hopital Saint-Andre, Bordeaux
  - APHM - Hospital Sainte Marguerite, Marseille
  - CHR Orleans, Orléans
  - Centre Hospitalier Annecy Genevois, Pringy
  - HU de Strasbourg - Nouvel Hopital Civil, Strasbourg

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Background] Priyanka Arora, Moti Ramgopal, Thomas CS Martin, Hui Liu, Jason T Hindman, Jason Okulicz, Dhananjay D Marathe, Samir Gupta Pharmacokinetics and Safety Data After Switching From Injectable CAB + RPV to Oral B/F/TAF 20th European AIDS Conference (EACS); October 15-18, 2025
- [Background] Samir Gupta, Thomas Martin, Cyril Gaultier, Alexandra Kissling, Kathleen Beusterien, Megan Chen, Megan Dunbar, Hui Liu, Brenda Ng, Moti Ramgopal Evaluation of Treatment Satisfaction and Experiences Among People With HIV When Switching to B/F/TAF From CAB + RPV: Results From the Phase 4 EMPOWER Study IDWeek; October 19-22, 2025; Atlanta, GA, USA
- [Background] Sharon Walmsley, Moti Ramgopal, Thomas Martin, Jason T Hindman, Hui Liu, Keith Aizen, Jason Okulicz, Samir Gupta A Phase 4 Study to Evaluate the Safety and Efficacy of Oral B/F/TAF After Discontinuing Injectable CAB + RPV IDWeek; October 19-22, 2025; Atlanta, GA, USA
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06104306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, France, and Canada.
Pre-assignment Details: 36 participants were screened.
Groups:
- Bictegravir/Emtricitabine/Tenofovir (B/F/TAF): Participants living with virologically suppressed HIV-1 infection who were unable/unwilling to continue on cabotegravir + rilpivirine (CAB + RPV) intramuscular (IM) injections or were wishing to switch to oral therapy, received a fixed dose combination of bictegravir/emtricitabine/tenofovir (B/F/TAF) 50/200/25 mg tablets orally, once daily for up to 24 weeks.
Period: Overall Study
Arm/Group | Bictegravir/Emtricitabine/Tenofovir (B/F/TAF)
Started | 33
Completed | 29
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Death | 1
Not completed — Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who have received at least 1 dose of the study drug (B/F/TAF).
Groups:
- B/F/TAF: Participants living with virologically suppressed HIV-1 infection who were unable/unwilling to continue on cabotegravir + rilpivirine (CAB + RPV) intramuscular (IM) injections or were wishing to switch to oral therapy, received a fixed dose combination of bictegravir/emtricitabine/tenofovir (B/F/TAF) 50/200/25 mg tablets orally, once daily for up to 24 weeks.
Arm/Group | B/F/TAF
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 18
  Race: Black or African American | 6
  Race: Not Collected | 4
  Race: Other or More Than One Race | 2
  Race: American Indian or Alaska Native | 1
  Race: Asian | 1
  Race: Native Hawaiian or Other Pacific Islander | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 20
  Ethnicity: Hispanic or Latino | 11
  Ethnicity: Not Collected | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27
  France | 4
  Canada | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment Emergent Grade 3 or 4 Drug-related Adverse Events Through Week 12 (Co-Primary Endpoint)
Description: Treatment emergent adverse events (TEAEs) were defined as any AE that began on or after the date of first dose of study drug up to the date of last dose of study drug plus 30 days or any AE leading to study drug discontinuation. The severity of AEs were be graded using the Division of AIDS (DAIDS) Toxicity Grading Scale.
  The DAIDS grading table provide an adverse events (AE) severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines:
  * Grade 1 indicates a mild event
  * Grade 2 indicates a moderate event
  * Grade 3 indicates a severe event
  * Grade 4 indicates a potentially life-threatening event
  * Grade 5 indicates death
Time Frame: Week 12
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- B/F/TAF: Participants living with virologically suppressed HIV-1 infection who were unable/unwilling to continue on CAB + RPV IM injections or were wishing to switch to oral therapy, received a fixed dose combination of B/F/TAF 50/200/25 mg tablets orally, once daily for up to 24 weeks.
Arm/Group | B/F/TAF
Number analyzed (Participants) | 33
percentage of participants | 0

2. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Grade 3 or 4 Laboratory Abnormalities Through Week 12 (Co-Primary Endpoint)
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any time after baseline up to and including the date of last dose of study drug plus 30 days.
  The DAIDS Toxicity Grading Scale, Version 2.1 was used to assign toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 included all values that did not meet the criteria for an abnormality of at least Grade 1. Grade 1 mild, Grade 2 moderate, Grade 3 severe, and Grade 4 potentially life-threatening.
Time Frame: Week 12
Population: Participants in the Safety Analysis Set with at least 1 postbaseline value for the test under evaluation, were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
percentage of participants | 3.1

3. Secondary Outcome: Plasma Concentrations of Cabotegravir (CAB), and Rilpivirine (RPV) at Day 1 (Predose)
Time Frame: Day 1 (Predose)
Population: CAB Pharmacokinetics (PK) Analysis Set and RPV PK Analysis Set included all enrolled participants who received at least 1 dose of study drug and CAB and RPV prior to joining the study, and had at least 1 nonmissing CAB and RPV concentration values reported by the PK laboratory tests. Participants in the CAB PK and RPV PK Analysis Sets with available data (samples collected as per the protocol) were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 29
ng/mL
  CAB | 1650 (1010)
  RPV | 68.3 (26.1)

4. Secondary Outcome: Plasma Concentration of Bictegravir (BIC), CAB, and RPV at Week 4
Time Frame: Week 4 (at trough and 2 hours postdose)
Population: BIC PK Analysis Set included all enrolled participants who received at least 1 dose of study drug and CAB and RPV prior to joining the study, and had at least 1 nonmissing BIC concentration value reported by the PK laboratory test. Participants in the BIC PK, CAB PK and RPV PK Analysis Sets with available data (samples collected as per the protocol) were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 25
ng/mL
  BIC, Trough: number analyzed (Participants) | 22
  BIC, Trough | 3590 (2030)
  BIC, 2 Hours Postdose | 6350 (2210)
  CAB, Trough: number analyzed (Participants) | 22
  CAB, Trough | 929 (739)
  CAB, 2 Hours Postdose | 975 (761)
  RPV, Trough: number analyzed (Participants) | 22
  RPV, Trough | 57.8 (20.8)
  RPV, 2 Hours Postdose | 55.7 (21.1)

5. Secondary Outcome: Plasma Concentration of BIC, CAB, and RPV at Week 12
Time Frame: Week 12 (at trough and 2 hours postdose)
Population: Participants in the BIC PK, CAB PK and RPV PK Analysis Sets with available data (samples collected as per the protocol) were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 24
ng/mL
  BIC, Trough: number analyzed (Participants) | 22
  BIC, Trough | 3850 (2550)
  BIC, 2 Hours Postdose | 6550 (2100)
  CAB, Trough: number analyzed (Participants) | 22
  CAB, Trough | 667 (982)
  CAB, 2 Hours Postdose | 647 (873)
  RPV, Trough: number analyzed (Participants) | 22
  RPV, Trough | 47.2 (22.4)
  RPV, 2 Hours Postdose | 45.4 (22.4)

6. Secondary Outcome: Plasma Concentration of BIC, CAB, and RPV at Week 24
Time Frame: Week 24 (at trough and 2 hours postdose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 20
ng/mL
  BIC, Trough: number analyzed (Participants) | 19
  BIC, Trough | 2820 (1530)
  BIC, 2 Hours Postdose | 6410 (1340)
  CAB, Trough: number analyzed (Participants) | 19
  CAB, Trough | NA (NA) — Data not available, as per the pre-specified analysis in the SAP, that data cannot be calculated where 1/3 participants had below the level of quantification (BLQ) concentrations.
  CAB, 2 Hours Postdose | NA (NA) — Data not available, as per the pre-specified analysis in the SAP, that data cannot be calculated where 1/3 participants had below the level of quantification (BLQ) concentrations.
  RPV, Trough: number analyzed (Participants) | 19
  RPV, Trough | 37.1 (22.3)
  RPV, 2 Hours Postdose | 33.1 (17.4)

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 12 as Determined by Missing = Excluded Approach
Description: This outcome measure analyzed using the Missing = Excluded (M = E) method. In this approach, all missing data were excluded in the analysis.
Time Frame: Week 12
Population: The Full Analysis Set included all enrolled participants who received at least 1 dose of the study drug (B/F/TAF). Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 30
percentage of participants | 0.0 [0.0 to 11.6]

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 24 as Determined by Missing = Excluded Approach
Description: as for outcome 7
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 29
percentage of participants | 0.0 [0.0 to 11.9]

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 12 as Determined by Discontinuation = Failure Approach
Description: This outcome measure was analyzed using the Discontinuation = Failure (D = F) method. In this approach, all discontinuation were treated as HIV-1 RNA >= 50 copies/mL (failure) in the analysis.
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 31
percentage of participants | 3.2 [0.1 to 16.7]

10. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 24 as Determined by Discontinuation = Failure Approach
Description: as for outcome 9
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
percentage of participants | 9.4 [2.0 to 25.0]

11. Secondary Outcome: Percentage of Participants With Discontinuation of B/F/TAF by Week 12
Time Frame: Up to 12 Weeks
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 33
percentage of participants | 3.0 [0.1 to 15.8]

12. Secondary Outcome: Percentage of Participants With Discontinuation of B/F/TAF by Week 24
Time Frame: Up to 24 Weeks
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 33
percentage of participants | 9.1 [1.9 to 24.3]

13. Secondary Outcome: Percentage of Participants Experiencing Treatment-emergent Grade 3 or 4 Laboratory Abnormalities Through Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: Participants in the Safety Analysis Set with at least 1 postbaseline value for the test under evaluation value were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
percentage of participants | 6.3

14. Secondary Outcome: HIV Treatment Satisfaction (HIVTSQc) Score at Week 4
Description: The HIVTSQc was a 1-12 items questionnaire. Each item was scored -3 to 3. The total score ranged from -33 to +33, based on 11 items. Higher the score, greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment. A score of 0 represented no change.
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
score on scale | 27 (9.0)

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 25 weeks; Adverse events: Up to 24 weeks plus 30 days
Description: All-cause mortality: The All Enrolled Analysis Set included all participants enrolled into the study after screening.
  Adverse events: The Safety Analysis Set included all enrolled participants who have received at least 1 dose of the study drug (B/F/TAF).
Arm/Group | B/F/TAF
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 10/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=33)
Abdominal pain upper (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=33)
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT06104306/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT06104306/SAP_001.pdf